CLINICAL TRIAL: NCT02214394
Title: Propofol in Exhaled Breath: Real-time Detection by Surface Acoustic Wave Sensors.
Brief Title: Detection of Propofol in Exhaled Breath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xhale Assurance (Industry)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20121475-00087006; 1R43GM090469-01A1 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propofol (Experimental): Subjects will be given Propofol during routine surgery and then using the SMART Device the breath will be captured and compared to blood plasma using High-performance liquid chromatography Analysis.
  Interventions: Other: High-performance liquid chromatography Analysis; Device: SMART Device

INTERVENTIONS:
Other: High-performance liquid chromatography Analysis — Blood samples will be collected for HPLC analysis to compare with the breath samples.
Device: SMART Device — Breath collection for GC-MS analysis to compare with Blood collection.
  Other Names: SMART Breath Based Monitor

SUMMARY:
This study involves the use of an experimental device which will measure how much propofol is present in your exhaled breath during surgery compared to how much is in your blood. The study results will look at whether the device is as accurate as conventional methods for measuring propofol levels during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old
* Healthy Male or Female
* BMI between 18.5 and 30.0
* Have a planned surgery or other medical procedure requiring anesthesia
* Physical status ASA I, II, or III

Exclusion Criteria:

* Known allergy to any component of propofol formulation components
* History of lung disease or tobacco use in the past 5 years
* Any finding not detailed above encountered on medical history or during screening physical and clinical laboratory examinations that, in the investigators judgment, might place the subject at unacceptable risk for injury during study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of propofol concentrations in exhaled breath to those in plasma | Sampling will occur every 2 minutes after anesthetic induction up to 10 minutes and then every 5 minutes thereafter up to 1 hour.
  Measure and compare propofol concentrations in exhaled breath to those in plasma in human patients anesthetized with propofol. Samples of the exhaled breath from patients will be monitored using the SAW Sensor and collected onto Tenax TA Tubes for analysis by Thermal Desorption GC/MS (using the method described by Grossher et al.)

CONTACTS AND LOCATIONS:
Overall Officials: Donn M Dennis, M.D., F.A.H.A., Study Director — Xhale, Inc.
Locations (1):
- University of Florida, Gainesville, Florida, United States